CLINICAL TRIAL: NCT04232475
Title: Effect of Stair Climbing and Descending on Postprandial Blood Glucose Following Mixed Meal
Brief Title: Effect of Stair Climbing and Descending on Postprandial Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeff Moore, Primary Investigator, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SCDPBG
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Postprandial Blood Glucose
MeSH Terms: interventions — Stair Climbing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Seated control
- 1 minute SCD (Experimental): 1 minute of stair climbing and descending
  Interventions: Other: 1 minute of stair climbing and descending
- 3 minute SCD (Experimental): 3 minute of stair climbing and descending
  Interventions: Other: 3 minute of stair climbing and descending
- 10 minute SCD (Experimental): 10 minute of stair climbing and descending
  Interventions: Other: 10 minute of stair climbing and descending

INTERVENTIONS:
Other: 1 minute of stair climbing and descending — 1 minute of stair climbing and descending
  Arms: 1 minute SCD
Other: 3 minute of stair climbing and descending — 3 minute of stair climbing and descending
  Arms: 3 minute SCD
Other: 10 minute of stair climbing and descending — 10 minute of stair climbing and descending
  Arms: 10 minute SCD

SUMMARY:
Determine effect of stair climbing and descending on postprandial blood glucose

DETAILED DESCRIPTION:
Determine effect of 1, 3, and 10 minutes of stair climbing and descending on postprandial blood glucose compared to seated control following consumption of mixed meal

ELIGIBILITY:
Inclusion Criteria:

* within specified age limit, ability to climb and descend stairs determined by ACSM's PAR-Q

Exclusion Criteria:

* diagnosis of diabetes or use of diabetic medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | 15 minutes
Postprandial blood glucose | 30 minutes
Postprandial blood glucose | 45 minutes
Postprandial blood glucose | 60 minutes
Postprandial Insulin | 15 minutes
Postprandial Insulin | 30 minutes
Postprandial Insulin | 45 minutes
Postprandial Insulin | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore JM, Salmons H, Vinoskey C, Hooshmand S, Kressler J. One minute of stair climbing and descending reduces postprandial insulin and glucose with 3-min improving insulin resistance following a mixed meal in young adults: A Randomized Controlled Crossover Trial. J Exerc Sci Fit. 2024 Jul;22(3):266-270. doi: 10.1016/j.jesf.2024.03.004. Epub 2024 Mar 18. PMID 38572086